CLINICAL TRIAL: NCT03165292
Title: An International Multicenter Phase II Randomised Trial Evaluating and Comparing Two Intensification Treatment Strategies for Metastatic Neuroblastoma Patients With a Poor Response to Induction Chemotherapy
Brief Title: Evaluation of 2 Intensification Treatment Strategies for Neuroblastoma Patients With a Poor Response to Induction
Acronym: VERITAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor has been notified of an interruption in the international supply, and there is a possibility that 131I-mlBG would be unavailable to patients randomised to arm A of the trial
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-003130-27; 2015/2294 (Other: CSET number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Very High Risk Neuroblastoma
MeSH Terms: interventions — 3-Iodobenzylguanidine; Topotecan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: High administered activity 131I-mIBG radiolabelled with iodine-131 and Topotecan (Experimental): The trial will evaluate two randomised arms. Each arm includes
  * three cycles of Temozolomide-Irinotecan, similar in both arms,
  * a specific consolidation course detailed hereinafter,
  * a BuMel sequence, followed by an ASCT, similar in both arms,
  * external radiotherapy as appropriate, and/or local surgery of the tumour residues as appropriate.
  Interventions: Radiation: mIBG; Drug: Topotecan; Procedure: Autologous stem cell transplant
- Arm B: High dose Thiotepa (Experimental): The trial will evaluate two randomised arms. Each arm includes
  * three cycles of Temozolomide-Irinotecan, similar in both arms,
  * a specific consolidation course detailed hereinafter,
  * a BuMel sequence, followed by an ASCT, similar in both arms,
  * external radiotherapy as appropriate, and/or local surgery of the tumour residues as appropriate.
  Interventions: Drug: Thiotepa; Procedure: Autologous stem cell transplant

INTERVENTIONS:
Radiation: mIBG — Day 1 131I-mIBG course 1: about 444MBq/kg with in vivo whole-body dosimetry Day 15 131I-mIBG course 2: the target is to deliver a combined whole-body radiation dose of 4 Gy
  Arms: Arm A: High administered activity 131I-mIBG radiolabelled with iodine-131 and Topotecan
Drug: Topotecan — Day 1-5 Topotecan 0.7 mg/m2 daily Day 15-19 Topotecan 0.7 mg/m2 daily
  Arms: Arm A: High administered activity 131I-mIBG radiolabelled with iodine-131 and Topotecan
Drug: Thiotepa — Day 1-3 Thiotepa
  Arms: Arm B: High dose Thiotepa
Procedure: Autologous stem cell transplant — ASCT as soon as radiation level allows it in ARM A

SUMMARY:
The main objective is to evaluate the efficacy of two intensified consolidation strategies in very-high risk neuroblastoma (VHR-NBL) patients in terms of event-free survival from randomisation date. This evaluation will follow a hierarchical testing procedure: each experimental treatment will be first evaluated as a single-arm phase 2 study, and in case of positive conclusion, the relative efficacy of both arms will then be evaluated comparatively.

DETAILED DESCRIPTION:
High-risk metastatic neuroblastoma is not cured by a single treatment. All patients who have become long-term survivors have received sequential treatments with various drugs.

For this reason, this trial does not compare two single treatments, but compares two sequential treatment strategies. In these two strategies, most of the components are evidence-based best practice, although the level of evidence supporting each component varies. There is one experimental component in each strategy. Indeed, none of these two treatment schedules can be considered as standard therapy, and none has been previously compared with any standard therapy in a randomised trial.

Although it might be considered that this trial should have a standard therapy arm as a comparator, analysis of patients treated in the SIOPEN HR NBL trial 1 who have failed to meet the R1 criteria has shown a wide heterogeneity of treatments. Therefore, there is no recognised or accepted standard treatment in this very high-risk patient group, and no guidelines exist for poor responders. Survival in this very high-risk group is currently very poor. Considering all these points, it is considered ethical to compare two experimental schedules without a standard comparator.

This trial compares two such strategies in a randomised way. Patients are eligible for entry into the trial if they fail to have an adequate response to induction and therefore cannot proceed directly within the high-risk study to BuMel PBSCR. Eligible patients will be randomised at that time point, even though further standard treatment will be administered before the randomised element, and there may be circumstances when an individual patient although randomised to a particular strategy, is unable to receive the randomised element of treatment. For example, if it proves impossible to perform an adequate PBSC harvest. All randomised patients will be analysed on an intention to treat basis.

Following randomisation, all patients will continue with standard dose chemotherapy with irinotecan and temozolomide for three courses to allow for PBSC harvest (it is not mandatory to have clear bone marrows before attempting a harvest) and to facilitate scheduling of the randomised element of the study which may necessitate referral to another centre.

The patients will then receive one of two investigational intensification therapies according to random allocation:

* high administered activity 131I-mIBG and topotecan and ASCR.
* high-dose thiotepa and ASCR Then all patients will proceed to second high-dose chemotherapy: BuMel and ASCR.

The intensified consolidation chemotherapy will be followed by external radiotherapy as appropriate, by local surgery of the tumour residues as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic neuroblastoma (NBL)
2. Patient previously treated within the ongoing High Risk Neuroblastoma SIOPEN study or treated with the current standard treatment for very high risk neuroblastoma off-trial
3. mIBG scintigraphy positive at diagnosis and after induction chemotherapy (pre BuMel evaluation).
4. Metastatic response after induction chemotherapy lower than the ongoing High Risk Neuroblastoma SIOPEN trial criteria to be eligible for High Dose Chemotherapy (metastatic response worse than partial response (< PR) or SIOPEN score > 3)
5. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of treatment. Sexually active patients must agree to use acceptable and appropriate contraception while on study drug and for one year after stopping the study drug. Acceptable contraception are defined in CTFG Guidelines "Recommendations related to contraception and pregnancy testing in clinical trials". Female patients who are lactating must agree to stop breast-feeding.
6. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local regional or national guidelines.
7. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.

Exclusion Criteria:

1. Parenchymal brain metastasis (even one)
2. Progressive disease at study entry
3. Previous high-dose therapy and Autologous Stem Cell Reinfusion
4. Performance status (Karnofsky, Lansky) <70%
5. Patient having received other therapy for cancer treatment than those allowed as per the ongoing High Risk Neuroblastoma SIOPEN trial or as defined in the future frontlines protocol (for HRNBL1 trial : after induction + 2 TVD)
6. Impaired organ function (liver, kidney, heart, lungs)

   * Shortening fraction <28%, or ejection fraction <55%, or clinical evidence of congestive heart failure or uncontrolled cardiac rhythm disturbance
   * Dyspnea at rest and/or pulse oxymetry <95% in air
   * ALT, Bilirubin > 2 ULN
   * Creatinine clearance and/or GFR < 60 ml/min/1.73m^2 and serum creatinine >/= 1.5 mg/dl
7. Any uncontrolled intercurrent illness or infection that in the investigator's opinion would impair study participation
8. Concomitant use with yellow fever vaccine and with live virus and bacterial vaccines
9. Patient allergic to peanut or soya
10. Chronic inflammatory bowel disease and/or bowel obstruction
11. Pregnant or breastfeeding women
12. Known hypersensitivity to the active substance or to any of the excipients of study drugs
13. Known hypersensitivity to dacarbazine
14. Concomitant use with St John's Wort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | From the randomisation into the VERITAS trial to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Valteau-Couanet, MD, PhD, Principal Investigator — Gustave roussy Paris, France
Locations (9):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - St. Anna Kinderspital GmbH, Vienna
- Gustave Roussy, Villejuif, Val De Marne, France
- Italy (3):
  - Meyer children's Hospita, Florence
  - Fondazione IRCCS Istituto nazionaleTumori, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
- Princess Maxima Center, Utrecht, Netherlands
- Spain (2):
  - Hospital Universitario Cruces, Cruces
  - Hospital Universitario y policnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR